CLINICAL TRIAL: NCT00483379
Title: An Exploratory, Open-Label Study of the Safety and Efficacy of High Dose or High Dosing Frequency Alglucosidase Alfa Treatment in Patients With Pompe Disease Who Do Not Have an Optimal Response to the Standard Dose Regimen
Brief Title: High Dose or High Dose Frequency Study of Alglucosidase Alfa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGLU03306
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Results first posted 2011-04-22 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-02

CONDITIONS: Pompe Disease; Glycogen Storage Disease Type II (GSD-II); Glycogenesis 2 Acid Maltase Deficiency
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- alglucosidase alfa 20 mg/kg every week (Experimental): Participants were treated with alglucosidase alfa 20 mg/kg every week for 52 weeks. This was the 'frequent dose' arm.
  Interventions: Biological: alglucosidase alfa
- alglucosidase alfa 40 mg/kg every other week (Experimental): Participants were treated with alglucosidase alfa 40 mg/kg every other week for 52 weeks. This was the 'high dose' arm.
  Interventions: Biological: alglucosidase alfa

INTERVENTIONS:
Biological: alglucosidase alfa — intravenous infusion
  Other Names: Recombinant human acid glucosidase; Myozyme

SUMMARY:
Pompe disease (also known as glycogen storage disease Type II) is caused by a deficiency of a critical enzyme in the body called acid alpha-glucosidase (GAA). Normally, GAA is used by the body's cells to break down glycogen (a stored form of sugar) within specialized structures called lysosomes. In patients with Pompe disease, an excessive amount of glycogen accumulates and is stored in various tissues, especially heart and skeletal muscle, which prevents their normal function. The objective of this exploratory study is to evaluate the safety and efficacy of alternative dosing regimens of alglucosidase alfa in patients with Pompe disease who have not demonstrated an optimal response to the standard dosing regimen of 20 mg/kg every other week after a minimum of 6 months treatment immediately prior to study entry.

ELIGIBILITY:
Inclusion Criteria:

* The patient or patient's legal guardian must provide signed, informed consent prior to performing any study-related procedures;
* The patient must have a clinical diagnosis of Pompe disease as defined by documented GAA deficiency in skin fibroblasts or blood;
* The patient must have been compliant with the standard dosing regimen of alglucosidase alfa (20 mg/kg every other week) for a minimum of 6 months immediately prior to study entry
* The patient must have clinical decline or sub-optimal improvement in at least one of the following parameters as compared to their condition prior to the beginning alglucosidase alfa treatment:

  1. Cardiac: Left Ventricular Mass (LVM) Z-score ≥6 or LVM index ≥150 g/m2 after a minimum of 6 months of regular treatment with alglucosidase alfa; OR
  2. Respiratory: New development of respiratory failure requiring the use of ventilatory assistance (invasive or non-invasive) after a minimum of 6 months of regular treatment with alglucosidase alfa. Ventilatory assistance must have been required for at least 4 weeks prior to study enrollment; OR
  3. Motor Skills:
* For patients ≤ 2 years of age at study entry, failure to acquire at least 2 new gross motor milestones after a minimum of 6 months of regular treatment with alglucosidase alfa; OR
* For patients > 2 years of age at study entry, worsening of proximal upper extremity muscle weakness as determined by the Investigator through loss of functional use of the upper extremities after a minimum of 6 months of regular treatment with alglucosidase alfa, OR
* For patients > 8 years of age at study entry, worsening of proximal upper extremity muscle weakness as determined by the Investigator through longitudinal assessments of manual muscle testing after a minimum of 6 months of regular treatment with alglucosidase alfa, OR
* For patients previously ambulatory, progression to use of an assistive device for ambulation due to worsening of proximal lower extremity muscle weakness after a minimum of 6 months of regular treatment with alglucosidase alfa.

Exclusion Criteria:

* For patients < 18 years of age, negative Cross-Reactive Immunologic Material (CRIM) assay result (added in protocol amendment #2);
* Any medical condition which, in the opinion of the Investigator, could interfere with treatment or evaluation of safety and/or efficacy of alglucosidase alfa;
* The patient is not currently receiving alglucosidase alfa;
* The patient has major congenital abnormality;
* The patient has used any investigational product (other than alglucosidase alfa in those regions where the product is not commercially available) within 30 days prior to study enrollment;
* The patient is pregnant or lactating.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-05; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (11):
- United States (9):
  - Birmingham, Alabama
  - Stanford, California
  - Washington D.C., District of Columbia
  - Chicago, Illinois
  - Kansas City, Kansas
  - Boston, Massachusetts
  - Grand Rapids, Michigan
  - Glenn Falls, New York
  - Durham, North Carolina
- Parkville Victoria, Australia
- Calgary, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fourteen participants were screened and enrolled; however, one withdrew before receiving any study infusions due to the burden of weekly trips to the medical center.
Period: Treatment Period
Arm/Group | Alglucosidase Alfa 20 mg/kg Every Week | Alglucosidase Alfa 40 mg/kg Every Other Week
Started | 6 | 7
Completed | 4 | 7
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Extension Period
Arm/Group | Alglucosidase Alfa 20 mg/kg Every Week | Alglucosidase Alfa 40 mg/kg Every Other Week
Started | 1 (Extension allowed late-onset participants access to treatment until commercially available.) | 2 (Extension allowed late-onset participants access to treatment until commercially available.)
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alglucosidase Alfa 20 mg/kg Every Week | Alglucosidase Alfa 40 mg/kg Every Other Week | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.3 (27.75) | 16.8 (15.56) | 19.8 (21.29)
Age, Customized [Number; unit: participants]
  <18 years | 4 | 5 | 9
  >= 18 and <=65 years | 2 | 2 | 4
  >65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Life-stage of Disease Onset [Number; unit: participants]
  Infantile-onset Pompe Disease | 4 | 5 | 9
  Late-onset Pompe Disease | 2 | 2 | 4
Parameter in Clinical Decline [Number; unit: participants] — Participant counts of the parameter in clinical decline (cardiac, respiratory or motor skills as compared to their condition prior to the beginning alglucosidase alfa treatment) for which participants were included in the study.
  participants
    Cardiac | 0 | 0 | 0
    Respiratory | 1 | 1 | 2
    Motor Skills | 5 | 6 | 11
Cross-Reactive Immunologic Material (CRIM) Assay Result [Number; unit: participants]
  Positive | 0 | 3 | 3
  Negative | 1 | 0 | 1
  Unknown | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Participants' Efficacy Response During the Treatment Period as Compared to Baseline for Participants With Respiratory Decline on Standard Treatment
Description: Participants were enrolled based on clinical decline or sub-optimal clinical response in cardiac, respiratory and/or motor function parameters pre-study while on standard treatment. Each participant was evaluated at Week 52 for change from baseline in the criteria that declined; respiratory decline as measured by change in ventilator use is summarized in this outcome. Ventilator use might have improved (less use of ventilator support), had no change, or worsened (more use of ventilator support). Each participant served as his or her own control.
Time Frame: Baseline, Week 52
Population: All participants who enrolled due to decline in respiratory function while on standard treatment.
Measure: Number; unit: participants
Arm/Group | Alglucosidase Alfa 20 mg/kg Every Week | Alglucosidase Alfa 40 mg/kg Every Other Week
Number analyzed (Participants) | 1 | 1
participants
  Improved | 0 | 0
  No change (on invasive ventilator for 24 hrs) | 0 | 1
  Worsened | 0 | 0
  Not evaluated | 1 | 0

2. Secondary Outcome: Baseline Values for Left Ventricular Mass (LVM) Z-Scores
Description: Z-Scores indicate the number of standard deviations (SD) from the mean in a normal distribution. Negative values indicate a smaller than mean LVM and values higher than 0 indicate a larger LVM than the mean. The normal range is -2 to 2 and greater than 2 may indicate left ventricular hypertrophy. The Z-scores for all parameters are calculated with reference to the normative data from the Children's Hospital, Boston, MA (Colan, 1992, J Am Coll Cardiol) based on the reference population with matched body surface area (BSA). Z-scores for LVM were provided by the central cardiologist.
Time Frame: Day 0
Population: Full analysis population of participants with LVM data
Measure: Median (Full Range); unit: Z-score
Arm/Group | Alglucosidase Alfa 20 mg/kg Every Week | Alglucosidase Alfa 40 mg/kg Every Other Week
Number analyzed (Participants) | 5 | 5
Z-score | 0.3 [-1.2 to 6.3] | -0.3 [-1.2 to 2.2]

3. Secondary Outcome: Change From Baseline in Left Ventricular Mass (LVM) Z-Score at Week 52
Description: Z-Scores indicate the number of standard deviations (SD) from the mean in a normal distribution. A negative change from baseline indicates a decrease and positive change from baseline an increase in LVM Z-score. The normal range is -2 to 2 and greater than 2 may indicate left ventricular hypertrophy. The Z-scores for all parameters are calculated with reference to the normative data from the Children's Hospital, Boston, MA (Colan, 1992, J Am Coll Cardiol) based on the reference population with matched body surface area (BSA). Z-scores for LVM were provided by the central cardiologist.
Time Frame: Baseline, Week 52
Population: Full analysis population of participants with LVM data at both timepoints
Measure: Median (Full Range); unit: Z-score
Arm/Group | Alglucosidase Alfa 20 mg/kg Every Week | Alglucosidase Alfa 40 mg/kg Every Other Week
Number analyzed (Participants) | 3 | 3
Z-score | 0.3 (1.04) [-0.8 to 1.2] | 0.4 (0.33) [-0.1 to 0.5]

4. Secondary Outcome: Baseline Values for Left Ventricular Mass Index (LVMI)
Description: Cardiac pathophysiology was assessed by a central cardiologist using left ventricular mass index (LVMI) measured by echocardiogram at Baseline. Left Ventricular Mass is adjusted to the participant's body surface area in the calculation of LVMI.
Time Frame: Day 0
Population: Full analysis population of participants with LVMI data
Measure: Median (Full Range); unit: g/m^2
Arm/Group | Alglucosidase Alfa 20 mg/kg Every Week | Alglucosidase Alfa 40 mg/kg Every Other Week
Number analyzed (Participants) | 5 | 5
g/m^2 | 62.1 [49.0 to 187.3] | 56.5 [45.4 to 73.1]

5. Secondary Outcome: Change From Baseline in Left Ventricular Mass Index (LVMI) at Week 52
Description: Cardiac pathophysiology was assessed by a central cardiologist using left ventricular mass index (LVMI) measured by echocardiogram at Baseline and after 12 months of treatment (Week 52). Left Ventricular Mass is adjusted to the participant's body surface area in the calculation of LVMI.
Time Frame: Baseline, Week 52
Population: Full analysis population of participants with LVMI data at both timepoints
Measure: Median (Full Range); unit: g/m^2
Arm/Group | Alglucosidase Alfa 20 mg/kg Every Week | Alglucosidase Alfa 40 mg/kg Every Other Week
Number analyzed (Participants) | 3 | 3
g/m^2 | 12.5 (14.44) [-10.9 to 15.5] | 4.0 (5.95) [-5.3 to 5.8]

6. Secondary Outcome: Change From Baseline in Ventilator Use at Last Assessment (Approximately Week 52)
Description: The change from baseline in ventilator use at the last assessment is summarized as improved (less use of ventilator support), no change, worsened (increased use of ventilator support), and did not use ventilator support.
Time Frame: Baseline, approximately Week 52
Population: Full analysis population. The participant in the worsened category died after week 52.
Measure: Number; unit: participants
Arm/Group | Alglucosidase Alfa 20 mg/kg Every Week | Alglucosidase Alfa 40 mg/kg Every Other Week
Number analyzed (Participants) | 6 | 7
participants
  Improved | 0 | 0
  No change | 2 | 3
  Worsened | 1 | 0
  Did not use ventilator | 3 | 4

7. Secondary Outcome: Change From Baseline in Body Strength Measured by the Manual Muscle Testing (MMT) Total Score at Week 52
Description: Body strength is measured by the MMT score on a scale of 0-10 with higher scores representing greater body strength.
Time Frame: Baseline, Week 52
Population: Full analysis population of participants >= 8 years old. Due to the age restriction and small study population, the number of participants analyzed is too small for results to be meaningful.
Arm/Group | Alglucosidase Alfa 20 mg/kg Every Week | Alglucosidase Alfa 40 mg/kg Every Other Week
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Baseline Values of Raw Scores for Gross Motor Function Measure 66 (GMFM-66) Results
Description: The Gross Motor Function Measure 66 contains sixty-six questions with a total raw score range of 0 - 198. Raw scores are derived from the following dimensions: Lying and rolling = 12; Sitting = 45; Crawling and kneeling = 30; Standing = 39; Walking, running and jumping = 72. Higher scores indicate better gross motor functions.
Time Frame: Day 0
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alglucosidase Alfa 20 mg/kg Every Week | Alglucosidase Alfa 40 mg/kg Every Other Week
Number analyzed (Participants) | 6 | 6
units on a scale | 65.0 (60.52) | 82.8 (84.00)

9. Secondary Outcome: Change From Baseline in Raw Scores for Gross Motor Function Measure 66 (GMFM-66) Results at Week 52
Description: as for outcome 8
Time Frame: Baseline, Week 52
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alglucosidase Alfa 20 mg/kg Every Week | Alglucosidase Alfa 40 mg/kg Every Other Week
Number analyzed (Participants) | 4 | 6
units on a scale | 6.0 (8.49) | 6.7 (6.12)

10. Secondary Outcome: Baseline Values in Mobility as Measured by the Pompe Pediatric Evaluation of Disability Inventory (Pompe PEDI)
Description: The Pompe PEDI is a disease specific version of the PEDI that was developed to assess functional capabilities and performance in children with Pompe disease from 2 months through adolescence. Baseline results for the mobility domain are reported. Scaled scores are used as an evaluative measure of change in performance over time with acquisition of new skills or new levels of independence. The range of scores is from 0-100 with scores near "0" reflecting low capability and scores near "100" reflecting high capability.
Time Frame: Day 0
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alglucosidase Alfa 20 mg/kg Every Week | Alglucosidase Alfa 40 mg/kg Every Other Week
Number analyzed (Participants) | 6 | 7
units on a scale | 38.3 (20.94) | 46.8 (21.26)

11. Secondary Outcome: Change From Baseline in Mobility as Measured by the Pompe Pediatric Evaluation of Disability Inventory (Pompe PEDI) at Week 52
Description: The Pompe PEDI is a disease specific version of the PEDI that was developed to assess functional capabilities and performance in children with Pompe disease from 2 months through adolescence. Change from baseline results for the mobility domain are reported. Scaled scores are used as an evaluative measure of change in performance over time with acquisition of new skills or new levels of independence. The range of scores is from 0-100 with scores near "0" reflecting low capability and scores near "100" reflecting high capability.
Time Frame: Baseline, Week 52
Population: Full analysis population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alglucosidase Alfa 20 mg/kg Every Week | Alglucosidase Alfa 40 mg/kg Every Other Week
Number analyzed (Participants) | 4 | 7
units on a scale | 0.6 (4.28) | 3.5 (3.84)

12. Secondary Outcome: Baseline Values for Normative Physical Component Summary of Medical Outcomes Study Short Form Health Survey (SF-36)
Description: Health related quality of life is measured using the Physical Component Summary (PCS) score of the Medical Outcomes Study (MOS) Short Form Health Survey (SF-36) for participants ≥14 years of age. SF-36 normative-based scoring has a mean of 50 and a standard deviation of 10. Higher scores represent better quality of life.
Time Frame: Day 0
Population: Full analysis population of participants >= 14 years old.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alglucosidase Alfa 20 mg/kg Every Week | Alglucosidase Alfa 40 mg/kg Every Other Week
Number analyzed (Participants) | 2 | 3
units on a scale | 31.3 (2.84) | 36.0 (9.33)

13. Secondary Outcome: Change From Baseline in Normative Physical Component Summary of Medical Outcomes Study Short Form Health Survey (SF-36) at Week 52
Description: as for outcome 12
Time Frame: Baseline, Week 52
Population: Full analysis population of participants >= 14 years old.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Alglucosidase Alfa 20 mg/kg Every Week | Alglucosidase Alfa 40 mg/kg Every Other Week
Number analyzed (Participants) | 1 | 3
units on a scale | 2.5 | 4.4 (11.24)

14. Primary Outcome: Participants' Efficacy Response During the Treatment Period as Compared to Baseline for Participants With Motor Function Decline on Standard Treatment
Description: Participants were enrolled based on clinical decline or sub-optimal clinical response in cardiac, respiratory and/or motor function parameters pre-study while on standard treatment. Each participant was evaluated at Week 52 for change from baseline in the criteria that declined; motor function decline primarily based on Gross Motor Function Measure 66 and Pompe Pediatric Evaluation of Disability Inventory results is summarized. Participants could gain motor function (improve), had no change (declined stopped), or continued loss (worsened). Each participant served as his or her own control.
Time Frame: Baseline, Week 52
Population: All participants who enrolled due to decline in motor function while on standard treatment.
Measure: Number; unit: participants
Arm/Group | Alglucosidase Alfa 20 mg/kg Every Week | Alglucosidase Alfa 40 mg/kg Every Other Week
Number analyzed (Participants) | 5 | 6
participants
  Gained gross or fine motor skills | 2 | 4
  No change | 1 | 2
  Continued motor loss | 1 | 0
  Not evaluated | 1 | 0

15. Primary Outcome: Summary of Participants Reporting Treatment-Emergent Adverse Events During the Treatment Period
Description: Overall safety summary of participants experiencing Adverse Events (AEs), Serious Adverse Events (SAEs), treatment-related AEs, and Infusion Associated Reactions (IARs). Summary is based on Treatment-emergent AEs (TEAEs), defined as AEs that occurred following the initiation of study treatment.
Time Frame: Day 1 up to Week 52
Population: Safety population comprised of all participants who received intervention.
Measure: Number; unit: participants
Arm/Group | Alglucosidase Alfa 20 mg/kg Every Week | Alglucosidase Alfa 40 mg/kg Every Other Week
Number analyzed (Participants) | 6 | 7
participants
  Participants with AEs | 6 | 7
  Related AEs | 0 | 2
  Not related AEs | 6 | 7
  Mild AEs | 6 | 6
  Moderate AEs | 3 | 2
  Severe AEs | 2 | 0
  AEs leading to discontinuation from study | 1 | 0
  Deaths | 1 | 0
  Infusion Associated Reactions | 0 | 2
  Serious AEs | 2 | 1

ADVERSE EVENTS:
Time Frame: Treatment period AEs were collected up to week 52. Extension period AEs were collected following completion of the treatment period until the product was commercially available (up to week 118).
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
  Events are listed independent of relationship to treatment reported.
Groups:
- Treatment: Alglucosidase Alfa 20 mg/kg Every Week: Participants were treated with alglucosidase alfa 20 mg/kg every week for 52 weeks. This was the 'frequent dose' arm.
- Treatment: Alglucosidase Alfa 40 mg/kg Every Other Week: Participants were treated with alglucosidase alfa 40 mg/kg every other week for 52 weeks. This was the 'high dose' arm.
- Extension: Alglucosidase Alfa 20 mg/kg Every Week; Extension: Alglucosidase Alfa 40 mg/kg Every Other Week: The extension period of the study allowed late-onset participants access to the same treatment they took in the treatment period until the product was commercially available.
Arm/Group | Treatment: Alglucosidase Alfa 20 mg/kg Every Week | Treatment: Alglucosidase Alfa 40 mg/kg Every Other Week | Extension: Alglucosidase Alfa 20 mg/kg Every Week | Extension: Alglucosidase Alfa 40 mg/kg Every Other Week
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/7 | 1/1 | 0/2
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 1/1 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment: Alglucosidase Alfa 20 mg/kg Every Week (N=6) | Treatment: Alglucosidase Alfa 40 mg/kg Every Other Week (N=7) | Extension: Alglucosidase Alfa 20 mg/kg Every Week (N=1) | Extension: Alglucosidase Alfa 40 mg/kg Every Other Week (N=2)
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment: Alglucosidase Alfa 20 mg/kg Every Week (N=6) | Treatment: Alglucosidase Alfa 40 mg/kg Every Other Week (N=7) | Extension: Alglucosidase Alfa 20 mg/kg Every Week (N=1) | Extension: Alglucosidase Alfa 40 mg/kg Every Other Week (N=2)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Right ventricular hypertrophy (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Amalgam tattoo (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Generalised oedema (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 2 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0 | 0
Pneumococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 2 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Aspiration tracheal abnormal (Investigations) | 0 | 1 | 0 | 0
Blood calcium increased (Investigations) | 1 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 1 | 0 | 0 | 0
Heart rate irregular (Investigations) | 1 | 0 | 0 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0 | 0 | 0
Protein urine present (Investigations) | 1 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Blood pressure fluctuation (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
This small exploratory study lacked a parallel control arm at the standard dose for a longer period; decline in respiratory or motor function prior to study was not collected systematically, thus change from baseline observations are inconclusive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI will delay submission of a publication until the earlier of; (i) publication of the multi-center data by Genzyme (ii)12-24 months after study completion or termination of the Study at all sites, or (iii) Genzyme notification that a publication will not occur. PI will send Genzyme a draft 60 days before publication. Genzyme can defer publication 90-120 days upon notifying PI that it will file a patent application on inventions contained in the draft.